CLINICAL TRIAL: NCT04393649
Title: First Level Socio-geriatric Evaluation in Period of Physical and Social Distancing in Frail Older Patients and Older Community Dwellers: ESOGER Databank
Brief Title: First Level Socio-geriatric Evaluation: ESOGER Databank
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Senior clinician researcher, Jewish General Hospital
Other Study IDs: MP-05-2021-2308
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: COVID; Social Isolation; Anxiety; Frailty
MeSH Terms: conditions — Social Isolation; Anxiety Disorders; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older patients / community dwellers: The inclusion criteria are:
  1. Older (i.e., 70-years-old and over) adults OR caregiver living at home with an adult answering to inclusion criteria
  2. Living and staying at home because of physical and social distancing
  3. Understanding and writing the different languages of the recruitment centre (i.e., French, English, Chinese.)
  4. Agree to participate in the study
  The exclusion criteria are:
  1. A concomitant participation to another medical trial
  2. Living in semi-autonomous residence or CHSLD
  Interventions: Other: ESOGER

INTERVENTIONS:
Other: ESOGER — Questionnaire

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an infectious disease. Physical distancing is one of the most effective ways to reduce the spread of COVID-19, but this key prevention intervention may have adverse consequences on older adults living at home. Screening older adults living at home and at risk for adverse consequences of physical and social distancing is, therefore, a priority in order to prevent their occurrence. ESOGER ("Evaluation Social et GERiatrique") is a clinical tool designed to: 1) screen the risk-levels for adverse consequences related to COVID-19 physical distancing and 2) to continue appropriate preventive interventions in older adults living at home including frail older patients and older community dwellers. Experience cumulated during the past two weeks revealed that ESOGER could be improved, in order to be more effective and efficient for the prevention of adverse consequences related to COVID-19 physical distancing. This improvement is based on two key components: 1) Comments of Montreal ESOGER users and 2) Analysis of data. Because at this time no information is saved and stored, there is a need to save and store ESOGER information and create the ESOGER databank.

ELIGIBILITY:
The inclusion criteria are:

1. Older (i.e., 70-years-old and over) adults OR caregiver living at home with an adult answering to inclusion criteria
2. Living and staying at home because of physical and social distancing
3. Understanding and writing the different languages of the recruitment centre (i.e., French, English, Chinese.)
4. Agree to participate in the study

The exclusion criteria are:

1. A concomitant participation to another medical trial
2. Living in semi-autonomous residence or CHSLD

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: All the older patients and community dwellers living at home in Montreal contacted by the researchers and corresponding to the criteria.
  The project is about a constitution of a databank.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2027-04-19 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
COVID-19 symptoms | 1 day
  presence or not of fever, cough and shortness of breath (binary question)
issues related to medication and food delivery and access to home care | 1 day
  presence or not of a rupture of access to food, medication and home care (binary question)
physical frailty | 1 day
  Questionnaire Emergency Room Evaluation and Recommandation (ER2), score from 0 = no risk of frailty to 14 = high risk of frailty)
psychological frailty | 1 day
  anxiety Verbal analogic scale, score from 0 = no anxiety to 10 = extremely anxious)

SECONDARY OUTCOMES:
Caregiver burden | 1 day
  Zarit scale, score from 0 = no caregiver burden to 16 = high caregiver burden)

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided